CLINICAL TRIAL: NCT06533202
Title: Study Protocol for a Randomised Controlled Trial: Effect of a Psycho-educational Intervention Programme for Comprehensive Preparation for Retirement and the New Phase of Life
Brief Title: Psycho-educational Intervention Programme for Comprehensive Preparation for Retirement: Study Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Sara Jiménez García-Tizón, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USAL
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Aging; Adaptation; Psychosocial Factors; Psychology; Older People; Retirement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The work of sequencing, randomisation, recruitment and allocation of the trial sample will be carried out by research staff who are not involved in the assessments or interventions of each group, thus avoiding any potential bias in the trial.
  Participants will also be blinded and will not know which group they have been allocated to and therefore which intervention they will receive. In order to minimise any contamination between groups, the assessment process will be carried out by external research staff who will perform the measurements and who have been previously trained and educated to avoid subjective bias in the process, as they will be unaware of the intervention group to which they have been assigned, thus masking the blinded assessment by third parties in the clinical trial. In addition, the researchers responsible for the statistical analysis of the trial will be blinded in order to increase the rigour of the trial process and thus the scientific quality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Programme (Active Comparator): Why: At the end of the baseline assessment, participants will receive instructions and recommendations to facilitate a positive and healthy transition to retirement, as part of an education programme. These will focus on the benefits of an active lifestyle and general guidelines to follow.
  What (materials): Instructions and recommendations for an education programme.
  What (procedures): Participants will receive instructions and recommendations on how to facilitate a positive and healthy transition to retirement as part of an education programme.
  How: The participants will receive the material individually at the commencement of the programme.
  When and for how long: The intervention consists of a single session and details of the time and duration will be provided to participants.
  Interventions: Behavioral: Education Programme
- Psychoeducational Programme (Experimental): Why: The programme is based on a psychoeducational intervention that aims to facilitate a positive and healthy transition into retirement.
  What (materials): projector, computer, screen, presentation of content, stationery, chairs, tables and self-recording of home tasks.
  What (procedures): Patients assigned to the experimental group will follow a psychoeducational programme structured and supervised at the University of Salamanca, consisting of a education programme combined with a psychoeducational programme.
  Who will carry out the interventions: The content is divided into six modules: (I) Introduction to retirement from a psychosocial approach, (II) Health and retirement, (III) Financial security and the process of successful retirement, (IV) Status and retirement, (V) Leisure and retirement, and (VI) My personal project (Table 1).
  When and for how long: Each participant will receive 4 sessions per month for 3 months, for a total of 12 sessions.
  Interventions: Behavioral: Psychoeducational Programme

INTERVENTIONS:
Behavioral: Psychoeducational Programme — The objective of this type of programme is to equip individuals with the knowledge and skills required to navigate the challenges and capitalise on the opportunities presented by retirement. In particular, the programme strives to enhance the quality of life and attitudes towards retirement, elevate levels of life satisfaction, psychological flexibility, perceived social support and general health, self-efficacy and self-regulation, and mitigate stereotypes associated with ageing.
  Arms: Psychoeducational Programme
Behavioral: Education Programme — At the end of the baseline assessment, participants will receive instructions and recommendations to facilitate a positive and healthy transition to retirement, as part of an education programme. These will focus on the benefits of an active lifestyle and general guidelines to follow.
  Arms: Education Programme

SUMMARY:
Background: The transition to retirement can be a challenging event, necessitating the adjustment of new routines, roles and expectations. Such modifications have the potential to impact the individual's quality of life and psychosocial well-being. t is of the utmost importance to develop intervention programmes that prepare people for retirement, with the objective of facilitating a positive and healthy transition.

Methods: A parallel randomised controlled clinical trial with two arms will be conducted. The study will be conducted at the Faculty of Psychology of the University of Salamanca (USAL) in Spain. The study will recruit individuals aged 60 years or older who are already retired or who will retire within the next five years. The participants will be divided into two groups: the intervention group (IG), which will undergo a comprehensive psychoeducational intervention programme, and the control group (CG), which will engage in a controlled follow-up. The programme will comprise 12 sessions over a period of three months. All participants will be assessed at the outset and conclusion of the study, as well as after three months, during which time data regarding their socio-demographic characteristics and responses to the following scales will be collected: The World Health Organization Quality of Life Measure - Brief Version (WHOQOL-BREF), the Retirement Attitudes Scale (EAJ), the Satisfaction With Life Scale (SWLS), the Questionnaire of Stereotypes towards Old Age (CENVE), the Acceptance and Action Questionnaire-II (AAQ-II), the MOS Questionnaire of Perceived Social Support (MOS), the General Health Questionnaire (GHQ), the Generalised Self-Efficacy Scale (EAG) and the Self-Regulation Scale (EAR).

Discussion: The objective of this study is to enhance the comprehension and implementation of intervention programmes in anticipation of retirement and the subsequent phase of life. To this end, a comprehensive psychoeducational intervention is proposed, with the aim of improving quality of life and attitudes towards retirement, increasing life satisfaction, psychological flexibility, perceived social support and general health, self-efficacy and self-regulation, and reducing stereotypes about ageing. The programme is designed to equip individuals with the skills and knowledge to navigate the challenges and opportunities associated with the transition to retirement.

ELIGIBILITY:
Inclusion Criteria:

* Be retired or nearing retirement (within 5 years)
* Be 60 years of age or older
* Voluntarily sign the consent form to participate
* Complete the initial assessment

Exclusion Criteria:

* No evidence of literacy difficulties or a significant deficit in language comprehension
* Not meet any of the inclusion criteria.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-09-09 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Measure - Brief Version (WHOQOL-BREF) | Baseline; up to 24 weeks; 3 months follow up
  Quality of life. The range of scores is from 26 to 100 points. The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
Retirement Attitudes Scale (EAJ) | Baseline; up to 24 weeks; 3 months follow up
  Attitudes towards retirement. The range of scores is from 20 to 140 points. The final scores indicate more negative attitudes the higher the value obtained.
Satisfaction With Life Scale (SWLS) | Baseline; up to 24 weeks; 3 months follow up
  Satisfaction with life. The range of scores is from 5 to 25 points. A higher score indicates that the person is generally satisfied with his/her life.
Questionnaire of Stereotypes towards Old Age (CENVE) | Baseline; up to 24 weeks; 3 months follow up
  Stereotypes about ageing. The range of score is from 5 to 20 points. High scores indicate a high degree of belief in negative stereotypes of ageing.
The acceptance and action questionnaire-II (AAQ-II) | Baseline; up to 24 weeks; 3 months follow up
  Psychological inflexibility. The range of score is from 7 to 49 points. High scores indicate more psychological inflexibility.
MOS Questionnaire of Perceived Social Support (MOS) | Baseline; up to 24 weeks; 3 months follow up
  Perceived social support. The overall scores range from 20 to 100 points. The higher the score, the more social support the individual perceives.
Goldberg General Health Questionnaire (GHQ) | Baseline; up to 24 weeks; 3 months follow up
  Perceived general health. The overall scores range from 0 to 36 points. Higher scores correspond to a higher level of perceived health.
Generalised Self-Efficacy Scale (EAG) | Baseline; up to 24 weeks; 3 months follow up
  Self-efficacy. Scores range from 10 to 40 points. Higher scores indicate higher levels of self-efficacy.
Self-Regulation Scale (EAR) | Baseline; up to 24 weeks; 3 months follow up
  Self-regulation. Scores range from 7 to 35 points. Higher scores on the scale indicate a greater ability to control attention in the pursuit of goals, while lower scores may suggest difficulties in maintaining focus and attention to goals.

CONTACTS AND LOCATIONS:
Locations (1):
- Castilla y León, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
They will be made available to researchers in the document repository "GREDOS" of the University of Salamanca, Spain.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available at the end of the study.
Access Criteria: Open access for researchers.
URL: http://gredos.usal.es/